CLINICAL TRIAL: NCT03654118
Title: Long-term Review of a Cohort of Arthroscopic Bankart Interventions
Acronym: ISIS-2017
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3025; 2017-A01665-48 (Other: Id-RCB)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Anterior Shoulder Instability
Keywords: Arthroscopy; Bankart; Shoulder; ISIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ISIS cohort: Patients operated between December 2007 and December 2008 for recurrent shoulder instability using the arthroscopic procedure (Arthroscopic Bankart) in the investigative centers and presenting at the time of indication for surgery an ISIS score ≤ 4 points
  Phone follow-up
  Interventions: Other: Phone follow-up

INTERVENTIONS:
Other: Phone follow-up — Through a short phone interview :
  * Determination of a complication (Infection, capsulitis, recurrence)
  * Determination of the Rowe score
  * Determination of the Walch-Duplay score

SUMMARY:
Recurrent instability is the most common chronic shoulder pathology of the young and athletic patient. It is a source of functional, sporting and professional disability, and a permanent apprehension to the use of the affected shoulder.

Surgical treatment has been proposed for a long time by the reintegration of the labrum (intervention of Bankart) then by the making of an osteo-muscular stop (intervention of Latarjet).

Like in many domains, surgical techniques have evaluated towards the search for endoscopic alternatives to open surgery, more deleterious.

Bankart's intervention has been performed arthroscopically since the 1980s and remains the majority intervention in the United States. However, its success rate never reached that of open techniques, Bankart and Latarjet. Surgeons therefore sought the predictors of these failures in order to define the limits of the indications for arthroscopic Bankart intervention.

The determination and use of the preoperative instability score (Instability Severity Index Score : ISIS) described by Balg and Boileau is one of the ways to clarify these indications.

The aim of this study is to prospectively establish the values of the ISIS score to obtain an acceptable recurrence rate of long-term instability

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient who already volunteered in a first ISIS study

Inclusion Criteria of the ISIS Study:

* Patients operated between December 2007 and December 2008 for recurrent shoulder instability, according to the arthroscopic procedure (Arthroscopic Bankart) in the investigative centers and presenting at the time of the indication of operation an ISIS score of ≤ 4 points (regardless of the positive criteria) (see Annex 2- ISIS score)
* Age> 16 years
* Supported by a joint arthroscopic technique completed.
* Patient not objecting to his participation in the study

Exclusion Criteria (same as those of the ISIS study)

* First dislocation or resumption of another technique at the time of indication for surgery
* Voluntary or multidirectional instability at the time of the indication of operation
* Painful shoulder without instability felt at the time of the operative indication
* Lesion of the cap (perioperative report)
* Humeral lesions Avulsion Gleno-humeral Ligament (per-operative finding)
* Unsuccessful technique
* Major benefiting from a legal protection measure (safeguard of justice, trusteeship, guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated between December 2007 and December 2008 for recurrent shoulder instability, according to the arthroscopic procedure (Arthroscopic Bankart)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
Number of instability recurrence after arthroscopic Bankart intervention | Through study completion, 2 months on average
  The rate of instability recurrence 9 years after an arthroscopic Bankart intervention, is derived from the patient's responses to the interview

SECONDARY OUTCOMES:
Predictive value of the ISIS score in the occurrence of recurrence of instability | Through study completion, 2 months on average

CONTACTS AND LOCATIONS:
Overall Officials: Hervé THOMAZEAU, MD, PhD, Study Director — Rennes University Hospital
Locations (11):
- France (11):
  - Clinique parc Rambot Provençale, Aix-en-Provence
  - Clinique Générale d'Annecy, Annecy
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Clinique du Cambresis, Cambrai
  - Clinique des Cèdres, Échirolles
  - Clinique François 1er, Le Havre
  - Clinique du Sport de Bordeaux-Mérignac, Mérignac
  - Hôpital Archet II, Nice
  - Hôpital Saint-Antoine / APHP, Paris
  - Clinique Turin, Paris
  - Centre Hospitalier Universitaire de RENNES, Rennes

IPD SHARING:
Plan to Share IPD: Undecided